CLINICAL TRIAL: NCT03943472
Title: A Phase I Clinical Trial of T-Cells Targeting B-Cell Maturation Antigen for Subjects With Relapsed/Refractory Multiple Myeloma
Brief Title: BCMA Chimeric Antigen Receptor Expressing T Cells Therapy for Relapsed/Refractory Multiple Myeloma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hrain Biotechnology Co., Ltd. (Industry)
Collaborators: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: anti-BCMA CART
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Multiple Myeloma
Keywords: BCMA; CAR-T; multiple myeloma; Relapsed /Refractory
MeSH Terms: conditions — Multiple Myeloma | interventions — fludarabine; Cyclophosphamide; Immune Checkpoint Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anti-BCMA CAR-T (Experimental): Administration of anti-BCMA CAR-T cells to patients with multiple myeloma
  Interventions: Biological: Anti-BCMA CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide
- anti-BCMA CAR-T+ Immune inhibitors (Experimental): Administration of anti-BCMA CAR-T cells + Immune inhibitors to patients with multiple myeloma
  Interventions: Biological: Anti-BCMA CAR-T cells; Drug: Fludarabine; Drug: Cyclophosphamide; Drug: Immune inhibitors

INTERVENTIONS:
Biological: Anti-BCMA CAR-T cells — Retroviral vector-transduced autologous T cells to express anti-BCMA CAR
Drug: Fludarabine — 30mg/m2/d
Drug: Cyclophosphamide — 300mg/m2/d
Drug: Immune inhibitors — Immune inhibitors
  Arms: anti-BCMA CAR-T+ Immune inhibitors

SUMMARY:
The goal of this clinical trial is to study the feasibility and efficacy of anti-B-Cell Maturation Antigen (BCMA) expressing T cells in treating patients with multiple myeloma.

DETAILED DESCRIPTION:
Participants with BCMA-positive relapsed/refractory multiple myeloma can participate if all eligibility criteria are met. Tests required to determine eligibility include disease assessments, a physical exam, Electrocardiograph, CT/MRI/PET, and blood draws. Participants receive chemotherapy prior to the infusion of BCMA CAR+ T cells. After the infusion, participants will be followed for side effects and effect of BCMA CAR+ T cells. Study procedures may be performed while hospitalized.

ELIGIBILITY:
Inclusion Criteria:

* Expected survival > 12 weeks
* Diagnosis of Multiple Myeloma by MWG criteria 20
* Patients previously received at least 3 different prior treatment regimens for multiple myeloma, including alkylating agent, protein inhibitors, and immunomodulator, and have disease progression in the past 60 days
* Important organs function enough to tolerate this therapy
* At least 90 days after stem cell transplantation
* Accessible to intravenous injection, and no white blood cell collection contraindications
* Sexually active patients must be willing to utilize one of the more effective birth control methods for 30 days after the CTL infusion. Male partner should use a condom
* Able to understand and sign the Informed Consent Document.

Exclusion Criteria:

* Patients with symptoms of central nervous system
* Patients with second malignancies in addition to multiple myeloma
* Active hepatitis B or C, HIV infections
* Any other active diseases could affect the enrollment of this trial
* Suffering severe cardiovascular or respiratory disease
* Poorly controlled hypertension
* Long term use of immunosuppressive agents after organ transplantation, except currently receiving or recently received glucocorticoid treatment
* A history of mental illness and poorly controlled
* Screening showing target cell transduction efficacy is lower than 30%, or T cell proliferation is not enough for infusion (less than 5 fold)
* Occurrence of unstable pulmonary embolism, deep vein thrombosis, or other major arterial/venous thromboembolic events 30 days prior to assignment
* Women of child-bearing potential who are pregnant or breastfeeding during therapy, or have a planned pregnancy with 2 months after therapy
* Women of child-bearing potential who are not willing to practice birth control from the time of enrollment on this study and for 2 months after receiving the preparative regimen. Women of child bearing potential must have a negative serum or urine pregnancy test performed within 48 hours before infusion
* Active systemic infections or uncontrolled infection within 14 days prior enrollment
* Subjects suffering disease affects the understanding of informed consent or complying with study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-07-08 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 5.0 | 6 months
  Safety measured by occurrence of study related adverse effects defined by NCI CTCAE 5.0

SECONDARY OUTCOMES:
Overall complete remission rate defined by the standard response criteria for malignant lymphoma for each arm | 8 weeks
  Overall complete remission rate defined by the standard response criteria for malignant lymphoma for each arm
Duration of CAR-positive T cells in circulation | 6 months
  Duration of CAR-positive T cells in circulation

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No